CLINICAL TRIAL: NCT04334226
Title: The Impact of Preoperative Urostomy Education on Patients and Families
Acronym: StomABC Impact
Status: Completed | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Elizabeth Wulff-Burchfield, MD, Assistant Professor, Medical Oncology, University of Kansas Medical Center
Other Study IDs: 145269
Record Dates: First submitted 2020-04-01; First posted 2020-04-06 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Bladder Cancer; Urostomy
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient and Caregiver Dyad: Individuals who participated in the Stoma Boot Camp study and their caregiver will form a dyad
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — Interviews will explore the patient's and caregiver's experiences and perceptions of ostomy surgery prior to the Bootcamp and after the Bootcamp from a physical, psychological, social, and spiritual perspective

SUMMARY:
This is an observational study utilizing a qualitative descriptive methodology with a thematic analysis approach to explore the impact of a preoperative educational intervention ("Stoma Bootcamp") on patients and their family/informal caregivers

DETAILED DESCRIPTION:
This study will utilize a qualitative descriptive methodology with a thematic analysis approach. Individual interviews will be held with bladder cancer and caregiver dyads who participated in the Stoma Bootcamp study. Interviews will explore the patient's and caregiver's experiences and perceptions of ostomy surgery prior to the Bootcamp and after the Bootcamp from a physical, psychological, social, and spiritual perspective. Semi-structured interview guides will be developed using Engel Biopsychosocial Model (BPS),5 one guide geared towards patients and the second toward caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age ≥ 18 years) patients who underwent radical cystectomy for bladder cancer at the University of Kansas Medical Center since 2016, AND
* Participated in the Stoma Bootcamp preoperative educational intervention, AND
* Identified an informal/family caregiver who participated in Stoma Bootcamp with them.
* Patient-caregiver dyads must both consent to participation

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent radical cystectomy for bladder cancer at the University of Kansas Medical Center and participated in Stoma Botcamp and their caregivers
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Impact of Stoma Bootcamp preoperative educational program on patients and caregivers | Interviews are expected to last 10-20 minutes and analysis expected to last approximately one year
  The research team will open code a subset of interviews, develop a codebook, and continue rounds of coding and discussion until consensus on code and definitions is reached. Once consensus is reached, all transcripts will be coded using the codebook, categories will be developed, and emergent themes will be assessed. Once themes are identified, they will be placed into a thematic map. Data will be analyzed until thematic saturation is reached

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Cancer Center, Westwood, Kansas, United States

IPD SHARING:
Plan to Share IPD: No